CLINICAL TRIAL: NCT04313049
Title: LARA: Use of JACO2 Controlled by Joystick or by Voice Control System, in Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 582
Record Dates: First submitted 2020-02-25; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Muscular Dystrophies
MeSH Terms: conditions — Muscular Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor control (Active Comparator)
  Interventions: Device: JACO2
- Vocal control (Experimental)
  Interventions: Device: JACO2; Device: VOCAL CONTROL

INTERVENTIONS:
Device: JACO2 — Performing tasks using joystick control
Device: VOCAL CONTROL — Performing tasks using vocal control
  Arms: Vocal control

SUMMARY:
As part of the EMPATIA @ Lecco project, task 2.9 and task 4.5 respectively provide for the refinement and testing of robotic solutions on the market oriented towards patient empowerment. Within the LARA project, the JACO2 mechanical arm (Kinova Technology, Montreal, QC, Canada), a medical device, which can perform some functions as if it were the subject's arm, will be tested. JACO2 can be controlled by joystick, supplied with the system, or by voice control system, developed by CNR-ITIA to allow use even for those with severe strength impairments. The trial will involve patients with Duchenne Muscular Dystrophy (DMD), Becker Muscular Dystrophy (BMD), Limb Girdle Muscular Dystrophy (LGMD), congenital and Facioscapulohumeral Muscular Dystrophy (FSH) over the age of 10 years. In literature of the last decade we find evidence of social and personal benefits deriving from the use of assistive mechanical arms in daily life activities by patients with disabilities due to neuromuscular diseases. The results indicate improved quality of life, greater self-esteem and greater integration into society. In addition to the benefits for the person, it has been shown that the introduction of assistive technologies in the life of patients can lead to potential savings on direct and indirect costs of National Health Services. Assistive robotic arms have a potential user base of approximately 150,000 people only in the United States of America. This population includes subjects who have partially lost the function of the upper limb due to degenerative diseases or because of spinal cord injuries or infantile cerebral palsy. The number of potential users could increase by improving the usability of these systems that, at the moment, still require a certain functionality of the upper limb, in general, and of the hand, in particular. It is in fact known that the introduction of assistive technologies in daily life is not limited so much by the fact that patients do not accept or profit from them, but rather by the actual possibility of using them effectively. Therefore, a customization of the functionality of the devices based on needs and wishes of the patients alongside an improvement in their usability would lead to an increase in potential users. It is for this reason that usability, together with safety, has become one of the most studied topics in assistive robotics. In the case of assistive robotic manipulators, usability problems often concern their control which, even today, takes place through the use of joysticks that require fine motor skills in the hand. In fact, being systems with multiple degrees of freedom, that is, equipped with different segments that can translate (or rotate) in different directions, different buttons are integrated in the control joysticks in addition to the classic lever with knob. From this emerges the need to develop alternative joystick control methods that do not involve the use of the hand.

ELIGIBILITY:
Inclusion Criteria:

* Availability by the patient and /or those who take care of him/her to sign the informed consent
* Defined diagnosis of Muscular Dystrophy (Duchenne, Becker, Limb Girdle type 2, Facioscapulohumeral and congenital)
* Use of the wheelchair as a mean of movement
* Weakness in the muscular districts of the shoulder girdle and of proximal upper limb detected by MRC scale (Medical Research Council) between 0 and 3
* Cognitive skills that allow understanding and management of robot
* Aged over 10 years

Exclusion Criteria:

* Presence of important comorbidities (epilepsy, 24/24 hours dependence on non-invasive or invasive ventilotherapy)
* Behavioral and psychiatric disorders (e.g., emotional problems, depression)

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Usability of the device (System Usability Scale) | immediately after application of the device
  The main outcome measure is the System Usability Scale (SUS), a validated questionnaire that measures the usability of a device, during a single experimental session, lasting no more than one hour.

SECONDARY OUTCOMES:
Execution Time | immediately after application of the device
  Measurements of the time for tasks execution through the single experimental session
Usefulness of the device (Likert scale) | immediately after application of the device
  An ad hoc questionnaire (with a Likert score from 0 to 5) for the subjective evaluation of the tasks for which the robot is useful through the single experimental session

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Eugenio Medea, Bosisio Parini, LC, Italy

IPD SHARING:
Plan to Share IPD: No